CLINICAL TRIAL: NCT05229016
Title: Priming Subjects to Influence Responses to Patient Reported Outcome Measures
Brief Title: Priming and Patient Reported Outcome Measures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Northwestern University (Other); Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AAAT8186
Record Dates: First submitted 2022-01-22; First posted 2022-02-08 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Patient Participation; PROM
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Intervention Model Description: Patients will be assigned randomly to complete one of six patient reported outcome measures.
  Prior to completion of the patient reported outcome measures, patients will be randomly assigned to one of three groups: Group A where patients will be asked to reflect on positive health-related experiences, Group B where patients will be asked to reflect on negative health-related experiences, Group C where patients will not be asked to reflect on health-related experiences (Control).
Who Masked: Participant
Masking Description: Participants are masked from knowing the purpose of the study's hypothesis, which is that patient-related factors may influence scores of patient related outcome measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (18):
- Positive health-related experiences and EQ-5D-5L (Experimental): Reflecting on positive health-related experiences EQ-5D-5L questionnaire
  Interventions: Behavioral: Reflection on health-related experiences
- Negative health-related experiences and EQ-5D-5L (Experimental): Reflecting on negative health-related experiences EQ-5D-5L questionnaire
  Interventions: Behavioral: Reflection on health-related experiences
- Control and EQ-5D-5L (No Intervention): No intervention/ control group EQ-5D-5L questionnaire
- Positive health-related experiences and PROMIS (Experimental): Reflecting on positive health-related experiences PROMIS Global health v1.2 questionnaire
  Interventions: Behavioral: Reflection on health-related experiences
- Negative health-related experiences and PROMIS (Experimental): Reflecting on negative health-related experiences PROMIS Global health v1.2 questionnaire
  Interventions: Behavioral: Reflection on health-related experiences
- Control and PROMIS (No Intervention): No intervention/ control group PROMIS Global health v1.2 questionnaire
- Positive health-related experiences and SF-36 (Experimental): Reflecting on positive health-related experiences SF-36 questionnaire
  Interventions: Behavioral: Reflection on health-related experiences
- Negative health-related experiences and SF-36 (Experimental): Reflecting on negative health-related experiences SF-36 questionnaire
  Interventions: Behavioral: Reflection on health-related experiences
- Control and SF-36 (No Intervention): No intervention/ control group SF-36 questionnaire
- Positive health-related experiences and SNOT-22 (Experimental): Reflecting on positive health-related experiences SNOT-22 questionnaire
  Interventions: Behavioral: Reflection on health-related experiences
- Negative health-related experiences and SNOT-22 (Experimental): Reflecting on negative health-related experiences SNOT-22 questionnaire
  Interventions: Behavioral: Reflection on health-related experiences
- Control and SNOT-22 (No Intervention): No intervention/ control group SNOT-22 questionnaire
- Positive health-related experiences and RSDI (Experimental): Reflecting on positive health-related experiences RSDI questionnaire
  Interventions: Behavioral: Reflection on health-related experiences
- Negative health-related experiences and RSDI (Experimental): Reflecting on negative health-related experiences RSDI questionnaire
  Interventions: Behavioral: Reflection on health-related experiences
- Control and RSDI (No Intervention): No intervention/ control group RSDI questionnaire
- Positive health-related experiences and mini-RQLQ (Experimental): Reflecting on positive health-related experiences Mini-RQLQ questionnaire
  Interventions: Behavioral: Reflection on health-related experiences
- Negative health-related experiences and mini-RQLQ (Experimental): Reflecting on negative health-related experiences Mini-RQLQ questionnaire
  Interventions: Behavioral: Reflection on health-related experiences
- Control and mini-RQLQ (No Intervention): No intervention/ control group Mini-RQLQ questionnaire

INTERVENTIONS:
Behavioral: Reflection on health-related experiences — This is a questionnaire that was designed to make the patient reflect on positive or negative health-related experiences.
  Arms: Negative health-related experiences and EQ-5D-5L; Negative health-related experiences and PROMIS; Negative health-related experiences and RSDI; Negative health-related experiences and SF-36; Negative health-related experiences and SNOT-22; Negative health-related experiences and mini-RQLQ; Positive health-related experiences and EQ-5D-5L; Positive health-related experiences and PROMIS; Positive health-related experiences and RSDI; Positive health-related experiences and SF-36; Positive health-related experiences and SNOT-22; Positive health-related experiences and mini-RQLQ

SUMMARY:
The objective of the study is to assess which health-related questionnaire is the most accurate and reliable.

The hypothesis is that some health-related questionnaires are more reliable than others.

DETAILED DESCRIPTION:
The objective of the study is to test the reliability of patient reported outcome measures, and their robustness to patient-related factors.

Patients will be randomly assigned to complete 1 of 6 patient reported outcome measures. Patients will either be asked to reflect on health-related experiences or not prior to completion of the questionnaire. Basic non-identifiable demographic information, and a brief medical questionnaire will follow completion of the patient reported outcome measure.

Results from each individual patient reported outcome measure will be compared.

ELIGIBILITY:
Inclusion Criteria:

18 years of age and older, living in the US, fluent written and spoken English, able to consent

Exclusion Criteria:

Any criteria that does not meet the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
EQ-5D-5L score | 15 minutes
  For the EQ-5D-5L, a scale of 1 to 5 with descriptors is used to score the domains of mobility, self-care, usual activities, pain/ discomfort and anxiety/ depression. A higher score represents a worse outcome.
PROMIS Global health v1.2 score | 15 minutes
  For the PROMIS Global Health v1.2, a score of 4 to 20 is calculated for the global physical health domain, and a score of 4 to 20 is calculated for the global mental health domain. A higher score represents a worse outcome.
SF-36 score | 15 minutes
  For the SF-36, a score of 0 to 100 is calculated for the domains of physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/ fatigue, emotional well-being, social functioning, pain, and general health. A higher score represents a more favorable outcome.
Sinonasal Outcomes Test (SNOT)-22 score | 15 minutes
  For the SNOT-22, a total score of 0 to 110 is calculated. The higher the score, the worse the outcome.
Rhinosinusitis Disability Index (RSDI) score | 15 minutes
  For the RSDI, a total score of 0 to 120 is calculated. The higher the score, the worse the outcome.
mini-RQLQ score | 15 minutes
  For the mini-RQLQ, a score 0 to 18 is calculated for the activities domain, 0 to 12 for the practical problems domain, 0 to 18 for the nose symptoms domain, 0 to 18 for the eye symptoms domain, and 0 to 18 for the other symptoms domain. A higher score represents a worse outcome.

SECONDARY OUTCOMES:
Present Mood Visual Analogue Scale | 15 minutes
  10 cm visual analogue scale to rate mood. The scale is between 0 and 10. A higher score represents a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: David Gudis, MD, Principal Investigator — Columbia University
Locations (1):
- New York Presbyterian Hospital- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
IPD will potentially be shared upon reasonable request